CLINICAL TRIAL: NCT01211795
Title: Phase III Double Blind Randomized Placebo Controlled Trial Using 20% Intra-Oral Ketoprofen Gel for Migraine Prevention.
Brief Title: Topical Intra-Oral Ketoprofen for Migraine Prevention
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Behar, Caren, M.D. (Individual)
Responsible Party: Caren Behar MD FACP, NYMC
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: IND 79,629
Record Dates: First submitted 2010-09-27; First posted 2010-09-30 (Estimated); Last update posted 2011-06-08 (Estimated); Status verified 2011-06

CONDITIONS: Migraine
Keywords: Migraine; Prevention; Treatment; Ketoprofen; Trigeminal nerve
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Topical Ketoprofen gel (Active Comparator)
  Interventions: Drug: topical intraoral ketoprofen gel
- Placebo gel (Placebo Comparator)
  Interventions: Other: Placebo Gel

INTERVENTIONS:
Drug: topical intraoral ketoprofen gel — 20% ketoprofen oral gel is applied once daily by cotton swab to a branch of the trigeminal nerve on the maxillary gingival mucosa above the 2nd and 3rd molars. The swab is held in place for 2 minutes at the same time once daily.
  Arms: Topical Ketoprofen gel
Other: Placebo Gel — An identical oral gel, without ketoprofen, or 'placebo gel' is applied using a cotton swab, once daily to a branch of the trigeminal nerve on the maxillary gingival mucosa. It is held in place for 2 minutes, once daily.
  Arms: Placebo gel

SUMMARY:
Intra-Oral Topical Ketoprofen gel, applied to a branch of the trigeminal nerve, has been shown to prevent migraines when used once daily for 3 months in open label studies. This is a randomized, double-blind, placebo controlled phase III prevention trial to determine safety and efficacy.

DETAILED DESCRIPTION:
This is a 4 month trial. During the first month, a prospective headache diary is maintained. Migraine frequency, severity (1-10), duration, and all headache medications are recorded.

Patients are then randomized to receive active gel or placebo gel in double blind fashion.

Gel is applied to the posterior maxilla once daily for 3 months. A daily headache diary, as outlined above, is maintained throughout the trial. Patients may continue to take other migraine medications, as needed. No other new migraine therapies may be started during the trial.

ELIGIBILITY:
Inclusion Criteria:

* IHS Migraine with or without aura
* 18 y.o. or older
* at least 4 migraines per month

Exclusion Criteria:

* pregnancy
* other headache conditions
* chronic daily headache
* allergy or sensitivity to NSAIDs other severe illnesses

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2009-10; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Change in number of migraine days per month | 3 months
  Number of migraine days per month will be compared before gel use and at the end of 3 months of use.

SECONDARY OUTCOMES:
Change in migraine severity | 3 month total
  Average migraine severity on a scale of 1-10, will be compared prior to gel use, and at the end of 3 months
Change in migraine duration | 3 months
  Average migraine duration will be compared prior to gel use, and at the end of 3 months
Change in headache medication use | 3 months
  Change in headache medication use will be compared prior to gel use, and at the end of 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Caren Behar, MD, Principal Investigator — New York Medical College
Locations (1):
- New York Medical College, Valhalla, New York, United States